CLINICAL TRIAL: NCT04554121
Title: Efficacy of Personalizing Cognitive Remediation for Schizophrenia by Targeting Impairments in Early Auditory Processing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Alice A. Medalia, PhD, Professor, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAU8479; 1R01MH123561-01 (NIH); 7982 (Other: New York State Psychiatric Institute Institutional Review Board)
Record Dates: First submitted 2020-09-14; First posted 2020-09-18 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Cognitive Remediation
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brain Basics (Experimental): Brain Basics is a cognitive remediation intervention that emphasizes training in early auditory processing.
  Interventions: Behavioral: Brain Basics
- Brain Training (Active Comparator): Brain Training is a cognitive remediation intervention that targets a range of cognitive abilities
  Interventions: Behavioral: Brain Training

INTERVENTIONS:
Behavioral: Brain Basics — Computer-based exercises targeting impairments in cognitive domains (sensory processing, processing speed, attention, working memory, memory) are paired with verbal discussions and group-based activities to strengthen metacognition and to bridge newly learned cognitive skills to everyday.
  life.
  Arms: Brain Basics
Behavioral: Brain Training — Computer-based exercises targeting impairments in cognitive domains (processing speed, attention, working memory, executive functions) are paired with verbal discussions and group-based activities to strengthen metacognition and to bridge newly learned cognitive skills to everyday life.
  Arms: Brain Training

SUMMARY:
The primary aim of this study is to provide confirmation that Cognitive Remediation (CR) for schizophrenia, when personalized based on pre-treatment assessment of early auditory processing ability, facilitates improved cognitive and functional outcomes. Additional aims of this study address the mechanisms of treatment effect. The study uses a repeated-measures randomized trial design.

Enrollment will be by invitation, open to individuals receiving services at select community behavioral health facilities where CR is offered. Clients who are eligible for the service, who agree to participate in research and who meet inclusion/exclusion criteria will be assessed on outcome measures and categorized via performance on the Tone Matching (TM) test, as EAP impaired (EAP-) or EAP intact (EAP+). Subsequently, EAP- and EAP+ subgroups will be randomized to either (1) Brain Basics (BB; n = 100), an EAP-enhanced CR approach or (2) Brain Training (BT; n = 100), a routine CR approach. Participants will be invited to participate in a second pre-treatment assessment to measure electrophysiologic responses to auditory stimuli. All participants will be scheduled to repeat outcome measure assessments after treatment and after a follow-up period. The EAP- group receiving BB will be invited to repeat electrophysiological paradigms post-treatment to investigate mechanisms of change related to the CR intervention. Verbal learning will be the primary outcome with functional capacity the secondary outcome. EEG is exploratory and will examine neurophysiologic markers of need for and response to EAP training.

DETAILED DESCRIPTION:
This personalized Cognitive Remediation (CR) confirmatory efficacy trial will be conducted at behavioral health facilities offering CR, located within the New York metropolitan area. Participants for this study will include adults diagnosed with schizophrenia or schizoaffective disorder, age 18-68, who have identified cognitive health as a pertinent treatment for recovery goal attainment and are seeking CR services. Individuals referred to CR may be referred for research by their treating clinician or may be self-referred. Consented individuals will receive a numeric study ID which will be used to de-identify all data collected for research.

Time 1 (baseline) outcomes assessments conducted by the research team include early auditory processing (EAP) ability, cognitive ability, and functioning. Participants will be classified as EAP impaired (EAP-) or EAP intact (EAP+). Following completion of Time 1 assessments, assignment to treatment condition will be stratified by EAP ability and randomized to Brain Basics (BB, n=100) or Brain Training (BT, n=100). Participants will be invited to participate in a separate EEG assessment of Mismatch Negativity (MMN).

CR will be conducted by trained clinicians at each performance site. CR will entail 30, 60-minute sessions administered two times a week (approximately 15 weeks). All participants will continue to receive recovery oriented therapeutic activities. Participants will be scheduled to repeat behavioral assessments at Time 2 (post-treatment) and Time 3 (follow-up) with a research team member who is blind to treatment group. The EAP- group receiving Brain Basics will also repeat EEG paradigms at Time 2 to explore mechanisms of change related to the CR intervention.

Verbal learning will be the primary outcome with functional capacity the secondary outcome. EEG is exploratory and will examine neurophysiologic markers of need for and response to EAP training. Mediation analysis will examine whether gains in cognition (verbal learning) mediate the gains in EAP and functioning. This will inform our understanding of EAP as the therapeutic change mechanism for about half of CR participants and confirm that EAP training need not be given to those CR participants with baseline intact EAP.

ELIGIBILITY:
Inclusion Criteria:

* A primary DSM-5 diagnosis of schizophrenia or schizoaffective disorder
* Psychiatrically stable, as defined by no changes in psychotropic medication or psychiatric hospitalization in the most recent 21 days
* English-speaking

Exclusion Criteria:

* Indications of Intellectual Disability as documented in medical history or measured by < 70 premorbid Full Scale IQ
* Documented auditory disorder or known visual impairment; presence of neurological conditions that are impacting brain and cognitive functioning
* Unremitted substance dependence within the past six months
* Participation in cognitive remediation in the 24 months prior

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2025-10-24 (Actual); Study Completion 2025-12-08 (Actual)

PRIMARY OUTCOMES:
Change in Verbal Learning | 15 weeks
  Verbal Learning is assessed with the MATRICS Consensus Cognitive Battery Verbal Learning Domain score. The primary outcome will be change in this score from pre to post treatment such that a higher value represents a better outcome.

SECONDARY OUTCOMES:
Change in Functional Capacity | 15 weeks
  Functional Capacity is assessed with the UCSD Performance Based Skills Assessment, Brief version. The secondary outcome will be change in the total score from pre to post treatment such that a higher value represents a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Medalia, Ph.D., Principal Investigator — Columbia University
Locations (9):
- United States (9):
  - Laurel House, Stamford, Connecticut
  - Williamsburg Clinic, Brooklyn, New York
  - Institute for Community Living, Brooklyn, New York
  - Heights Hill Clinic, Brooklyn, New York
  - Mapleton Mental Health Services, Brooklyn, New York
  - The Bridge, Inc., New York, New York
  - Manhattan Psychiatric Center 125th Street Clinic, New York, New York
  - Rockland Psychiatric Center, Orangeburg, New York
  - Pibly Residential Programs Inc., The Bronx, New York

IPD SHARING:
Plan to Share IPD: Yes
Raw data will be made available for research to investigators working under a Federal Wide Assurance who meet security measures and data use agreement criteria associated with public repositories including the National Database for Clinical Trials related to Mental Illness (NDCT). Data will include baseline demographic data, and baseline and post raw data derived from primary and secondary outcome measures.
Time Frame: A list of all data expected to be collected in the project will be submitted by January 2021. Subsequently, descriptive and raw data will be submitted on a semi-annual basis. Unpublished de-identified data will be submitted prior to study completion and will be shared within one year after project completion, or when the data are published, whichever is earlier.
Access Criteria: Data in NIH repositories may be accessed through the NIH Data Access Committee which reviews data access and submission requests.